CLINICAL TRIAL: NCT05458947
Title: A Prospective Analysis of Physical Therapy Wound Care Modalities in Patients With Spinal Cord Injury
Brief Title: Physical Therapy Wound Care Modalities in Patients With Spinal Cord Injury (SCI)
Acronym: (SCI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00085228
Record Dates: First submitted 2022-07-06; First posted 2022-07-14 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-04

CONDITIONS: Spinal Cord Injuries; Pressure Injuries
Keywords: Wound Care; Physical Therapy; Pulsed wound irrigation; Electrical stimulation
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer | interventions — Electric Stimulation

STUDY DESIGN:
Intervention Model Description: To examine the effects of PT wound care modalities (PWI + ES, PWI only, and ES only) on wound healing in patients with SCI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- pulsed wound irrigation (PWI) (Experimental): The necrotic wound is irrigated with normal saline (0.9%) with an 8-12 pounds per square inch pressure (PSI) to provide a mechanical force to loosen necrotic tissue for wound healing
  Interventions: Procedure: pulsed wound irrigation (PWI)
- electrical stimulation (ES) (Experimental): ES works to promote the migration of cells based on natural cell polarity known as galvanotaxis, enhancing and mimicking the natural current of injury. By recreating the natural electrical fields of the skin, ES attracts immune cells vital to healing to wound to facilitate wound closure
  Interventions: Procedure: electrical stimulation (ES)
- electrical stimulation (ES) and pulsed wound irrigation (PWI) (Experimental): The necrotic wound is irrigated with normal saline (0.9%) with an 8-12 pounds per square inch pressure (PSI) to provide a mechanical force to loosen necrotic tissue for wound healing and ES to promote the migration of cells based on natural cell polarity known as galvanotaxis, enhancing and mimicking the natural current of injury. By recreating the natural electrical fields of the skin, ES attracts immune cells vital to healing to wound to facilitate wound closure
  Interventions: Procedure: electrical stimulation (ES) and pulsed wound irrigation (PWI)

INTERVENTIONS:
Procedure: pulsed wound irrigation (PWI) — necrotic wound is irrigated with normal saline (0.9%) with an 8-12 pounds per square inch pressure (PSI) to provide a mechanical force to loosen necrotic tissue for wound healing
  Arms: pulsed wound irrigation (PWI)
Procedure: electrical stimulation (ES) — high volt pulsed current (HVPC) is most effective in wound healing while decreasing risk of adverse skin reactions or mild burns under the electrodes
  Arms: electrical stimulation (ES)
Procedure: electrical stimulation (ES) and pulsed wound irrigation (PWI) — necrotic wound is irrigated with normal saline (0.9%) with an 8-12 pounds per square inch pressure (PSI) to provide a mechanical force to loosen necrotic tissue for wound healing and high volt pulsed current (HVPC) is most effective in wound healing while decreasing risk of adverse skin reactions or mild burns under the electrodes
  Arms: electrical stimulation (ES) and pulsed wound irrigation (PWI)

SUMMARY:
To examine the effects of Physical Therapist (PT) wound care modalities (pulsed wound irrigation (PWI) + electrical stimulation (ES), PWI only, and ES only) on wound healing in patients with spinal cord injuries (SCI).

DETAILED DESCRIPTION:
It is hypothesized that PWI + ES will demonstrate the greatest rate of wound healing due to the combined effect of these treatments, which positively impact several aspects of the wound healing cascade. It is hypothesized that all patients will demonstrate improved quality of life from receiving wound care treatments by Physical Therapists due to individualized education and treatments which engage patients in their wound healing process and promote self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled at inpatient rehabilitation at Carolinas Rehabilitation Charlotte
* Diagnosis of spinal cord injury and concomitant pressure injury to sacrum or ischium
* Agreeable to wound care treatment by Physical Therapist (PT)
* Able to perform informed consent
* Over 18 years of age
* Physician order for PT wound care evaluation and treatment
* Bates-Jensen Wound Assessment Tool (BWAT) >31 on initial evaluation

Exclusion Criteria:

* Pain which limits ability to tolerate wound care treatments
* Unable to perform informed consent
* Pregnancy
* Bates-Jensen Wound Assessment Tool (BWAT) <30 on initial evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Bates-Jensen Wound Assessment Tool (BWAT) score | Baseline
  15-item objective measure designed to assess wound status and track healing - related to healing on a 1 (healed) to 5 (severe) scale to create a summative score between 13-65 with lower scores indicating progression towards healing
Bates-Jensen Wound Assessment Tool (BWAT) score | Week 1
  15-item objective measure designed to assess wound status and track healing - related to healing on a 1 (healed) to 5 (severe) scale to create a summative score between 13-65 with lower scores indicating progression towards healing
Bates-Jensen Wound Assessment Tool (BWAT) score | Year 1
  15-item objective measure designed to assess wound status and track healing - related to healing on a 1 (healed) to 5 (severe) scale to create a summative score between 13-65 with lower scores indicating progression towards healing

SECONDARY OUTCOMES:
Change in The Spinal Cord Injury Quality of Life measurement system (SCI-QOL) Short Form Score | Baseline and Year 1
  measures health-related quality of life specific to patients with Spinal Cord Injuries (SCI) - Higher scores indicate worse functioning quality of life related to pressure injuries, while lower scores indicate fewer impairments

CONTACTS AND LOCATIONS:
Overall Officials: Erin Weeks, PT,DPT, CWS, Principal Investigator — Carolinas Rehabilitation
Locations (1):
- Carolinas Rehabilitation, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No